CLINICAL TRIAL: NCT03497026
Title: A Single-Center, Prospective, Single Arm Study to Evaluate the Performance of the Auris Robotic Endoscopy System for Bronchoscopic Procedures
Brief Title: Auris Robotic Endoscopy System for Bronchoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Mutual Termination
Sponsor: Auris Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DD082015
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Robotic Bronchoscopy (Experimental): Robotic bronchoscopy with Robotic Bronchoscopy Platform
  Interventions: Device: Robotic Bronchoscopy Platform

INTERVENTIONS:
Device: Robotic Bronchoscopy Platform — Eligible patients will undergo the robotic bronchoscopy for evaluation of suspected lung nodules.
  Other Names: The Monarch Platform

SUMMARY:
In this study, the performance related to the use of the novel Robotic Endoscopy Platform during bronchoscopic procedures will be evaluated.

DETAILED DESCRIPTION:
The early and accurate diagnosis of lung cancer is critical. However, many peripheral lung lesions are beyond the reach of conventional bronchoscopes. Additionally, alternative techniques, such as CT-guided or surgical biopsy, can carry increased risks to the patient. Diagnostic yield of flexible bronchoscopy is limited by its inability to guide biopsy instruments directly to the lesion. Varying technologies have been proposed to guide endobronchial biopsies, such as electromagnetic navigation, endobronchial ultrasound (EBUS) and computed tomography fluoroscopy. However, the correlation of real-time guidance and the ability to precisely direct a biopsy instrument is critical to biopsy success.

In this study , the novel Robotic Endoscopy Platform and its accessories will be used to provide bronchoscopic visualization of and access to patient airways for diagnostic procedures. Commercially available biopsy instruments will be used to acquire tissue for diagnostic purposes.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age;
2. Capable and willing to give informed consent;
3. Acceptable candidate for an elective, non-emergent bronchoscopic procedure;
4. Solid peripheral lung lesions suspected of malignancy, between 1.5-7cm in size identified on thin slice CT scan with 30 days of the intended bronchoscopy

Exclusion Criteria:

1. Medical contraindication to bronchoscopy;
2. Ground glass opacity lesions on pre-procedure CT
3. Participation in any other clinical trial 30 days before and throughout the duration of the study;
4. Uncontrolled or irreversible coagulopathy;
5. Female subjects who are pregnant or nursing or those of child-bearing potential refusing a pregnancy test;
6. CT scan done over a month before the bronchoscopy procedure.

Intra-Procedure Exclusion Criteria: Any presenting condition discovered intra-procedurally that in the opinion of the investigator would make participating in this study not in the patient's best interest.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Krishna, MD, Principal Investigator — El Camino Hospital
Locations (2):
- United States (2):
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation Mountain View Center, Mountain View, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robotic Bronchoscopy
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robotic Bronchoscopy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed the Intended Bronchoscopic Procedure With the Robotic Endoscopy Platform
Description: Completion of the intended bronchoscopic procedure is defined by the ability to acquire tissue with biopsy tools.
Time Frame: During the procedure, up to 2 hours
Population: due to termination after 4 subjects enrolled, no statistical analyses would have been performed or would be considered scientifically appropriate.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Bronchoscopy
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: from enrollment through patient follow-up; 6 weeks
Arm/Group | Robotic Bronchoscopy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Bronchoscopy (N=4)
hospital admission for planned surgery (Respiratory, thoracic and mediastinal disorders) | 2 (2) — planned hospital admission
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Bronchoscopy (N=4)
coughing (Respiratory, thoracic and mediastinal disorders) | 4 (4)
sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study mutually terminated, no data analyzed

DOCUMENTS (1):
  • Study Protocol (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT03497026/Prot_001.pdf